CLINICAL TRIAL: NCT03230214
Title: Effect of Bacterial Translocation on Haemodynamic and Coagulation Parameters During a Liver Transplantation
Brief Title: Effect of Bacterial Translocation on Haemodynamic and Coagulation Parameters During Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Heba Moharem, assisstant lecturer, Alexandria University
Other Study IDs: 020583
Record Dates: First submitted 2017-07-20; First posted 2017-07-26 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Effect of Bacterial Translocation
MeSH Terms: interventions — Bacterial Translocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- DNA positive patients: patients who have bacterial DNA in their samples
  Interventions: Diagnostic Test: PCR for bacterial translocation
- DNA negative patients: patients who do not have bacterial DNA in their samples
  Interventions: Diagnostic Test: PCR for bacterial translocation

INTERVENTIONS:
Diagnostic Test: PCR for bacterial translocation — samples taken from the blood and ascites of patients to search for bacterial DNA

SUMMARY:
The present study is to demonstrate the effect of the presence of bacterial translocation detected by bacterial deoxyribonucleic acid (bactDNA) in blood and ascites using the polymerase chain reaction (PCR) on some haemodynamic and coagulation parameters during a liver transplant procedure.

ELIGIBILITY:
Inclusion Criteria:

• patients with liver failure undergoing liver transplantation

Exclusion Criteria:

* Age less than 18 years;
* Active overt infection;
* Patients on oral or systemic anticoagulation or with known coagulopathic disorders apart from those caused by liver failure (eg.: Protein C or S deficiency, congenital platelet disorders and congenital coagulation disorders…etc);
* Patients undergoing re-transplantation.

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult patients with grade C liver cirrhosis with liver failure undergoing liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
change in the mean arterial blood pressure | at the beginning of surgery then 15 nim after dissection then 15 min after the anhepatic phase then 15 min at the reperfusion phase
antifactor X activity | at the beginning of surgery
change in the heart rate | at the beginning of surgery then 15 nim after dissection then 15 min after the anhepatic phase then 15 min at the reperfusion phase
change in the cardiac output | at the beginning of surgery then 15 nim after dissection then 15 min after the anhepatic phase then 15 min at the reperfusion phase

CONTACTS AND LOCATIONS:
Overall Officials: ahmed mukhtar, MD, Study Director — Cairo University
Locations (1):
- Elmoasah Hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Moharem HA, Fetouh FA, Darwish HM, Ghaith D, Elayashy M, Hussein A, Elsayed R, Khalil MM, Abdelaal A, ElMeteini M, Mukhtar A. Effects of bacterial translocation on hemodynamic and coagulation parameters during living-donor liver transplant. BMC Anesthesiol. 2018 Apr 25;18(1):46. doi: 10.1186/s12871-018-0507-7. PMID 29699477